CLINICAL TRIAL: NCT01980966
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Study in Healthy Volunteers to Evaluate the Efficacy and Safety of MHAA4549A in an Influenza Challenge Model
Brief Title: A Study of MHAA4549A in Healthy Volunteers in an Influenza Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GV28985; 2013-001983-52 (EudraCT Number)
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- MHAA4549A (Experimental)
  Interventions: Drug: MHAA549A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Tamiflu (Active Comparator)
  Interventions: Drug: oseltamivir [Tamiflu]

INTERVENTIONS:
Drug: MHAA549A — IV dose
  Arms: MHAA4549A
Drug: Placebo — IV dose
  Arms: Placebo
Drug: oseltamivir [Tamiflu] — Orally b.i.d, 5 days
  Arms: Tamiflu

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of MHAA4549A in healthy volunteers in an influenza challenge model. Subjects will be intranasally oculated with the challenge virus and will be randomly assigned to receive a intravenous dose of either MHAA4549A or placebo. In the stage 5 cohort, subjects will be randomly assigned to receive doses of MHAA4549A or placebo or Tamiflu (oseltamivir) orally twice daily for 5 days. All subjects in all cohorts may take Tamiflu twice daily from Day 7 to Day 11.

ELIGIBILITY:
Inclusion Criteria:

* In good health with no history of major medical conditions from medical history, physical examination and routine laboratory tests
* Male subjects and women of child-bearing potential must use effective contraception as defined by protocol, starting at entry to quarantine and continuing until Day 120 follow-up visit
* Sero-suitable for challenge virus

Exclusion Criteria:

* Women who have been pregnant within 6 months prior to the study, or who have been breastfeeding within 3 months prior to the study, or who have a positive pregnancy test at any point in the study
* Any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinological, haematological, hepatic, immunological, metabolic, urological, neurological, psychiatric, renal, and/or other major disease or malignancy, as judged by the CI
* Abnormal pulmonary function evidenced by clinically significant abnormalities in spirometry
* History of asthma, COPD, pulmonary hypertension, reactive airway disease, or chronic lung disease of any etiology. A history of childhood asthma before the age of 12 is acceptable provided the subject is asymptomatic without treatment.
* History suggestive of respiratory infection within 14 days prior to admission to the unit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2014-06-19 (Actual); Study Completion 2014-06-19 (Actual)

PRIMARY OUTCOMES:
Viral area under the concentration-time curve (AUC) of nasopharyngeal viral load by quantitative Polymerase Chain Reaction (qPCR) | 8 days

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 120 days
Safety: Change in lung function | from pre-challenge to Day 29
Safety: Incidence of anti-therapeutic antibodies (ATAs) | 120 days
Pharmacokinetics: Area under the concentration-time curve | 8 days
AUC of nasopharyngeal viral load, as measured by cell culture | 8 days
Peak viral load (qPCR and cell culture) | 8 days
Duration of viral shedding | 8 days
Duration of Grade 2 or worse symptoms (from first occurrence of any Grade >2 symptom to last occurrence of any Grade >2 symptom) | 8 days
Peak/AUC of composite symptoms | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Retroscreen Ltd, London, United Kingdom

REFERENCES:
- [Derived] McBride JM, Lim JJ, Burgess T, Deng R, Derby MA, Maia M, Horn P, Siddiqui O, Sheinson D, Chen-Harris H, Newton EM, Fillos D, Nazzal D, Rosenberger CM, Ohlson MB, Lambkin-Williams R, Fathi H, Harris JM, Tavel JA. Phase 2 Randomized Trial of the Safety and Efficacy of MHAA4549A, a Broadly Neutralizing Monoclonal Antibody, in a Human Influenza A Virus Challenge Model. Antimicrob Agents Chemother. 2017 Oct 24;61(11):e01154-17. doi: 10.1128/AAC.01154-17. Print 2017 Nov. PMID 28807912
- [Derived] Deng R, Lee AP, Maia M, Lim JJ, Burgess T, Horn P, Derby MA, Newton E, Tavel JA, Hanley WD. Pharmacokinetics of MHAA4549A, an Anti-Influenza A Monoclonal Antibody, in Healthy Subjects Challenged with Influenza A Virus in a Phase IIa Randomized Trial. Clin Pharmacokinet. 2018 Mar;57(3):367-377. doi: 10.1007/s40262-017-0564-y. PMID 28639229